CLINICAL TRIAL: NCT06663111
Title: Rituximab and Ocrelizumab in Serum With Multiple Sclerosis (ROS-MS)
Brief Title: Rituximab and Ocrelizumab in Serum With Multiple Sclerosis
Acronym: ROS-MS
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 228768
Record Dates: First submitted 2022-01-31; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Blood samples for PK — Blood sampled for pharmacokinetic study
Other: Blood samples for PK — Blood samples before, shortly after infusion of already assigned/ongoing treatment as well as after 2, 4, 8, 12, 24 weeks for serum conc. measurements.

SUMMARY:
ROS-MS is a clinical pharmacological substudy to the OVERLORD-MS study (NCT04578639), designed to examine the possibilities of personalized treatment with rituximab and ocrelizumab in patients with relapsing-remitting multiple sclerosis.

DETAILED DESCRIPTION:
OVERLORD-MS is a 30 months prospective randomized double blinded multicenter non-inferiority study. The objective of OVERLORD-MS is to demonstrate if rituximab is non-inferior to ocrelizumab with regards to efficacy and safety in treatment naïve patients with relapsing-remitting multiple sclerosis (RRMS), diagnosed within the last 12 months.

In the patients enrolled in the clinical pharmacological substudy ROS-MS the serum concentrations of rituximab and ocrelizumab will be quantified using liquid chromatography tandem mass spectrometry (LC MS/MS) at predefined points during the dosing interval. Relevant biochemical parameters will also be analyzed in these samples.

Based on these measurements, the investigators will examine correlations between serum concentrations, biochemical parameters and the clinical outcomes in the OVERLORD-MS study. The objective is to evaluate whether clinical pharmacological tools, such as therapeutic drug monitoring (TDM) and pharmacokinetic pharmacodynamic models (PK-PD models), may be of value in the personalization of treatment with rituximab and ocrelizumab in patients with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Included in OVERLORD-MS (NCT04578639)
* Willing to attend laboratory for blood sample collection at scheduled time points

Exclusion criteria:

* Not willing to attend laboratory for blood sample collection at scheduled time points

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In OVERLORD-MS, treatment-naïve male and female patients aged 18-60 years, with newly diagnosed multiple sclerosis, are randomized 2:1 to treatment with rituximab or ocrelizumab. In the sub-study ROS-MS, patients are recruited from the patients included i OVERLORD-MS.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum drug concentration measured using liquid chromatography tandem mass spectrometry (LC-MS/MS) | Up to 24 weeks (during one cycle of treatment, injection of rituximab or ocrelizumab is scheduled every 6 months)
  The serum concentration of rituximab or ocrelizumab after drug infusion (maximum serum concentration (Cmax)) and 2, 4, 8, 12, 24 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Trond T. Serkland, M.D., Principal Investigator — Haukeland University Hospital; Silje Skrede, M.D., PhD, Study Director — University of Bergen
Locations (1):
- Haukeland University Hospital, Deparment of medical biochemistry and pharmacology, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No